CLINICAL TRIAL: NCT04378439
Title: Harnessing the Power of Peer Navigation and mHealth to Reduce Health Disparities in Appalachia
Brief Title: Appalachian Partnership to Reduce Disparities (Aim 2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00065116
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: HIV/AIDS; STI; HCV
Keywords: PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): 7 community health leaders; 56 social network members
  Interventions: Behavioral: Peer Navigation; Behavioral: mHealth
- delayed-intervention (Active Comparator): 7 community health leaders; 56 social network members
  Interventions: Behavioral: Peer Navigation; Behavioral: mHealth

INTERVENTIONS:
Behavioral: Peer Navigation — First, as health advisors, community health leaders will raise awareness of HIV, STIs, and HCV and local prevention and care services and help social network members access services. Thus, the community health leader will describe to the process for HCV testing, and how providers are required to maintain confidentiality. As opinion leaders, community health leaders will reframe health-compromising and bolster health-promoting norms and expectations about testing and use of other prevention and care services.
  Each community health leader will also conduct formal in-person group activities with their social network members. Our partnership decided that each community health leader will also hold at least 4 formal group sessions during the 12 months of intervention
Behavioral: mHealth — In addition to in-person individual and group activities, community health leaders will use mHealth platforms preferred by each social network member (i.e., Facebook , Instagram, testing, and/or GPS-based mobile apps) to communicate with them during the intervention. They will use social media to plan activities and to support use of needed prevention and care services. For example, when planning a group activity (described above), the community health leader will use social media to remind social network members about the activity and help them problem solve barriers to attending. A community health leader and social network member may also communicate "in-real-time" via social media about the process of participating in a syringe services program or accessing PrEP.

SUMMARY:
By combining two strategies (i.e., peer navigation and mHealth) into a complete, culturally compatible, bilingual intervention to increase the use of needed HIV, STI, and HCV prevention and care services among racially/ethnically diverse GBMSM and transgender women in rural Appalachia.

Study Investigators anticipate that participants in the intervention group, relative to counterparts in the delayed-intervention group, will demonstrate increased HIV, STI, and HCV testing.

DETAILED DESCRIPTION:
This CBPR study will advance prevention science and practice through testing an innovative intervention to promote and support the use of needed HIV, STI, and HCV prevention and care services among GBMSM and transgender women; and developing priorities and recommendations to improve their health that will be disseminated to inform public health practice, research, and policy. By integrating peer navigation and mHealth strategies, the proposed study provides a unique opportunity to improve health among vulnerable, hidden, and neglected populations living in rural Appalachia. Findings from this research may inform strategies and approaches to address other health disparities in other rural populations.

ELIGIBILITY:
Inclusion Criteria:

* reside in one of the rural Appalachian catchment countiesreside in one of the rural Appalachian catchment counties
* be ≥18 years of age
* report being assigned male sex at birth and having had sex with at least 1 man in past 12 months
* provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — GBMSM (Gay, Bisexual, Men who have sex with men)
Enrollment: 141 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have Human Immunodeficiency Virus (HIV) testing | baseline
Number of participants who have Sexually Transmitted Infection (STI) testing | baseline
Number of participants who have Hepatitis C Virus (HCV) testing | baseline
Number of participants who have HIV testing | immediate post-intervention (12 months post-baseline)
Number of participants who have STI testing | immediate post-intervention (12 months post-baseline)
Number of participants who have HCV testing | immediate post-intervention (12 months post-baseline)
Number of participants who have HIV testing | 12-month follow-up (24 months post-baseline)
Number of participants who have STI testing | 12-month follow-up (24 months post-baseline)
Number of participants who have HCV testing | 12-month follow-up (24 months post-baseline)

SECONDARY OUTCOMES:
Number of participants who use prevention--Pre-exposure prophylaxis (PrEP) | baseline, immediate post-intervention (12 months post-baseline), and 12-month follow-up (24 months post-baseline).
Number of participants who use prevention--syringe services | baseline, immediate post-intervention (12 months post-baseline), and 12-month follow-up (24 months post-baseline).
Number of participants who use HIV care services | baseline, immediate post-intervention (12 months post-baseline), and 12-month follow-up (24 months post-baseline).
  Measured through self-report and medical chart abstraction
Number of participants who use STI treatment services | baseline, immediate post-intervention (12 months post-baseline), and 12-month follow-up (24 months post-baseline).
  Measured through self-report and medical chart abstraction
Number of participants who use HCV treatment services | baseline, immediate post-intervention (12 months post-baseline), and 12-month follow-up (24 months post-baseline).
  Measured through self-report and medical chart abstraction
Number of participants who use gender-affirming care services | baseline, immediate post-intervention (12 months post-baseline), and 12-month follow-up (24 months post-baseline).
  Measured through self-report and medical chart abstraction

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Rhodes, Ph.D, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No